CLINICAL TRIAL: NCT05084846
Title: Influenza and the Heart: An Investigation Into the Acute and Lasting Cardiac Effects of Influenza Infection
Brief Title: InFLUenza and the HEART An Investigation Into the Acute and Lasting Cardiac Effects of Influenza Infection
Acronym: FluHeart
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Tor Biering-Sørensen, Associate Professor and Research Director, University Hospital, Gentofte, Copenhagen
Other Study IDs: H-21011835
Record Dates: First submitted 2021-10-06; First posted 2021-10-20 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Influenza; Cardiovascular Complication
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
"Influenza and the Heart: An investigation into the acute and lasting cardiac effects of influenza infection" the investigators aim to assess the mechanisms for cardiovascular disease in patients suffering an acute influenza infection. The project will be carried out by creating a prospective clinical cohort study of consecutive patients hospitalized at Herlev & Gentofte University Hospital with a laboratory confirmed influenza.

ELIGIBILITY:
Inclusion Criteria:

* All patients hospitalized at Herlev & Gentofte University Hospital with a laboratory-confirmed diagnosis of influenza
* > 18 years of age

Exclusion Criteria:

* Persons not able to cooperate
* Persons unable to understand and sign "informed consent"
* Pregnancy
* Persons simultaneously positive with COVID-19

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients with laboratory confirmed influenza
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients developing cardiovascular complications | 3 years
  Including new-onset heart failure, worsening of current heart failure, acute myocardial infarction, and cardiac arrest
Number of patients developing in-hospital mortality | 3 years
Rate of cardiac dysfunction | 3 years
  Defined by impaired echocardiographic parameters and elevated cardiac biomarkers - NT
  - pro
  - BNP annd hs
  - TNT
Prevalence of elevated biomarkers of infection/inflammation | 3 years
  Prevalence of elevated biomarkers of infection/inflammation and it association with cardiac dysfunction
Rate of pulmonary embolisms diagnosed with CT thorax angiography | 3 years

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Herlev & Gentofte Hospital, Copenhagen
  - Cardiovascular Non-Invasive Imaging Research Laboratory, department of Cardiology, Herlev & Gentofte Hospital, Hellerup